CLINICAL TRIAL: NCT03482583
Title: Implementation Strategies to Improve Tobacco Treatment for UF Health Cancer Center Patients
Brief Title: Tobacco Use Treatment in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702115 -A; OCR17294 (Other: UF OnCore)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Smoking, Cigarette
Keywords: Smoking, Cancer, Treatment
MeSH Terms: conditions — Cigarette Smoking; Smoking; Neoplasms | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cognitive Behavior Therapy with NRT (Other): Cognitive Behavior Therapy (CBT) will be provided by a certified tobacco treatment specialist (CTTS) using vidyo, a HIPAA-compliant video based platform. Participants in this arm, if interested will be provided a 2 week supply of nicotine replacement therapy (NRT). The intervention in this arm would be NRT along with the CBT counseling.
  Interventions: Drug: Nicotine Replacement Therapy
- Referral to Area Health Education Center (Other): The Area Health Education Center (AHEC) is a locally available tobacco cessation program aimed at strengthening the capacity of Florida's healthcare system to deliver effective evidence based tobacco use treatment, and prevention services throughout the state. The intervention is education on the health effects related to tobacco use, and benefits of quitting and what to expect when quitting. A tobacco cessation specialist of trained facilitator guides participants as they identify triggers and withdrawal symptoms, and discuss ways to cope with them. The program offers free nicotine replacement therapy, educational materials, goodies for their quit day and follow up support.
  Interventions: Other: Referral to AHEC/Quitline
- Referral to Qutiline (Other): Quitline is a local program in the state where smokers can call a toll free number to talk to coach who can help them quit. There is also an option of online program if they prefer to engage in online help to quit tobacco use.
  The intervention in this arm is counseling support by phone or online with an option of Nicotine replacement therapy. If participants prefer this option, our nurse will refer them to locally available quitline service using EPIC.
  Interventions: Other: Referral to AHEC/Quitline

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — Participants in CBT group will also be offered Nicotine Replacement Therapy if they are interested. NRT is the same regimen followed in AHEC and Quitline. In addition, weekly counseling will be provided to the participants remotely via vidyo, a video based platform.
  Other Names: Nicotine Patch
  Arms: Cognitive Behavior Therapy with NRT
Other: Referral to AHEC/Quitline — Participants will be referred to local AHEC/Quitline for treatment
  Arms: Referral to Area Health Education Center; Referral to Qutiline

SUMMARY:
Tobacco use among cancer survivors reduces the effectiveness of cancer treatments, increases the risk for additional primary cancers, and increases mortality. Implementation of tobacco treatment for cancer patients is challenging, but may be improved substantially with clinically-efficient and sustainable solutions to accurately identify tobacco users, direct them to evidence-based treatment, and provide demonstrable outcomes for stakeholders.

At UF Health Cancer Center (UFHCC), patient access and utilization of tobacco use treatment are sub optimal. Further, UFHCC has a largely rural catchment area with a high burden of tobacco-related disease and mortality. To address this research-to-practice gap using a mixed-methods approach to assess the relevant contextual factors at UFHCC and evaluate the feasibility of implementing a multi-level intervention to increase tobacco treatment utilization and improve health outcomes.

This study uses a mixed methods approach and will inform the design of a pragmatic clinical trial to improve the delivery of tobacco use treatment services to cancer patients. Guided by a conceptual model that emphasizes patient, provider, and organizational characteristics, the study team will identify factors that influence the implementation process at the UFHCC. The ultimate goal of the proposed research is to provide new knowledge to facilitate the widespread adoption, implementation, and dissemination and sustained utilization of evidence-based tobacco use treatments in cancer care settings.

DETAILED DESCRIPTION:
Study Design: This study uses a mixed methods approach and will inform the design of a pragmatic clinical trial to improve the delivery of tobacco use treatment services to cancer patients.

Study Setting: The pilot study will be conducted at the UF Health Medical Oncology and Ear, Nose & Throat (ENT) clinics. Smoking is the leading cause of head and neck cancers, and almost one-third of patients continue to smoke after their head and neck cancer diagnosis, making this a priority population for intervention.

Population: UF Health cancer patients ≥18 yrs old who are current smokers and smartphone users; for mCBT, the investigators will also ensure CO breath sample >5 parts per million (ppm). Patients with unstable medical or psychiatric illness or use disorder for illicit drugs will be excluded.

Procedures: The investigators will request Epic access to identify potential subjects and schedule recruitment during clinic hours. Research assistants (RAs) will be at the Medical Oncology and ENT clinics to meet with eligible patients during their visit. RAs will approach eligible patients at checkout after they are introduced by someone who has a clinical relationship with the patient. Following screening and brief counseling by the provider, RAs will offer eligible patients the 3 TUT options (i.e., AHEC, Quitline, or mCBT), obtain informed consent using REDCap (eConsent) or a paper consent (if desired by the patient), administer the Patient Exit Interview (PEI) in REDCap, and arrange a follow-up phone interview. Patients who choose AHEC/Quitline will be referred by a nurse using Epic. Those choosing mCBT will be trained on the use of Vidyo and the iCOTM Smokelyzer® by the RA, and follow-up will be arranged with a CTTS counselor.

Participants in mCBT will meet with a trained certified tobacco treatment counselor on Vidyo for 30 minutes, once a week, for 6 weeks. The counselor will cover topics that include addiction, withdrawal, dealing with triggers, overcoming cravings, and relapse prevention. At enrollment, investigators will offer mCBT participants-if interested-a 2-week supply of nicotine replacement therapy (NRT). The 2-week supply of NRT is consistent with what is offered to participants at AHEC and the Quitline. Participants who smoke less than 10 cigarettes per day will receive 14 mg of NRT, and those who smoke more than 10 cigarettes per day will receive 21 mg of NRT. Medical clearance from the provider will be obtained prior to NRT administration. At the end of the study (week 12), participants (all participants in mCBT and a random sample of patients referred to AHEC/Quitline) will complete the follow-up telephone interview. At the end of the study, participants (AHEC/Quitline & mCBT) may also provide a saliva sample to test their cotinine level; this process will be remotely monitored via Vidyo for participants in mCBT and participants in AHEC/Quitline will be encouraged to contact study staff to answer any questions they may have. Evaluation tools also consist of Patient Exit Interviews and Telephone Survey to be administered among research participants.

Analysis Plan: All data collected will be entered in a REDCap database. The primary analysis will be the estimation of rates/means, with 95% CIs. To demonstrate the feasibility of the 3 implementation strategies, investigators will measure reach as the number of smokers visiting the 2 clinics who are referred to any TUT (i.e., AHEC/Quitline/mCBT) divided by the total number of smokers visiting the clinics. For each TUT, investigators will calculate enrollment as the total number of smokers who enroll in a given treatment divided by the total number of referred smokers; investigators will compare the rates of patients selecting into each of the 3 TUT programs. Investigators will assess TUT completion as the number of enrolled smokers who complete the program. Investigators will also evaluate acceptability using TAQ. As secondary outcomes, investigators will measure prolonged abstinence at week 12 and the change (baseline to week 12) in past-7-day point prevalence (all programs), as well as CO-verified abstinence at weeks 6 &12 (mCBT only). CO levels will also be modeled across time (weeks 1, 6, 12) to assess for reductions over time via linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* UF Health cancer patients, 18 years and older, who are current smokers.

Exclusion Criteria:

* Patients with unstable medical or psychiatric illness or
* Patients with a use disorder for illicit drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi G. Salloum, PhD, MBA, Principal Investigator — University of Florida
Locations (5):
- United States (5):
  - UF Ear Nose and Throat (ENT), Gainesville, Florida
  - UF Health at the University of Florida, Gainesville, Florida
  - UF Health Medical Oncology, Gainesville, Florida
  - UF Health Radiation Oncology, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Referral to Qutiline: Quitline is a local program in the state where smokers can call a toll free number to talk to coach who can help them quit. There is also an option of online program if they prefer to engage in online help to quit tobacco use.
  The intervention in this arm is counseling support by phone or online with an option of Nicotine replacement therapy. If participants prefer this option, our nurse will refer them to locally available quitline service using EPIC.
  Referral to AHEC/Quitline: Participants will be referred to local AHEC/Quitline for treatment
Period: Overall Study
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline
Started | 37 | 14 | 39
Completed | 12 | 5 | 18
Not Completed | 25 | 9 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline | Total
Number analyzed (Participants) | 37 | 14 | 39 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.1) | 57.3 (6.9) | 60.6 (1.2) | 58.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 19 | 50
  Male | 16 | 4 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 36 | 13 | 39 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 9 | 30 | 68
  Black/African American | 5 | 4 | 8 | 17
  Other | 4 | 3 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 14 | 39 | 90
Rurality [Count of Participants; unit: Participants]
  Urban | 26 | 8 | 28 | 62
  Rural | 11 | 6 | 11 | 28
Cigarette Smoking Frequency [Count of Participants; unit: Participants]
  Every Day | 34 | 13 | 30 | 77
  Some Days | 3 | 0 | 7 | 10
  Declined to answer | 0 | 1 | 2 | 3
E-Cigarette Use Frequency [Count of Participants; unit: Participants]
  Every Day | 4 | 1 | 1 | 6
  Some Days | 6 | 1 | 10 | 17
  Not at All | 27 | 11 | 27 | 65
  Declined to Answer | 0 | 1 | 1 | 2
Cigarettes/Day [Mean (Standard Deviation); unit: Cigarettes/day] | 13.8 (12.1) | 20.1 (15.1) | 12.3 (8.5) | 14.2 (11.5)
Age of Smoking Initiation [Mean (Standard Deviation); unit: years] | 16.2 (6.4) | 21.0 (8.1) | 18.9 (6.2) | 17.0 (8.0)
Patient Exit Interview (PEI) [Mean (Standard Deviation); unit: units on a scale] — The Patient Exit Interview (PEI) is a 10-item patient-reported assessment of provider delivery of tobacco counseling, with each item scored as a 0 or a 1. The PEI composite score (range 0-10) is the sum of intervention steps each patient reports that the provider implemented, with higher scores indicating greater implementation of tobacco counseling. Assessment completed after recruitment and before intervention.
  units on a scale | 7.7 (2.6) | 6.9 (2.9) | 7.2 (2.9) | 7.4 (2.7)
Cancer Diagnosis [Count of Participants; unit: Participants]
  Past Week | 2 | 1 | 2 | 5
  Past Month | 5 | 0 | 4 | 9
  Past 1-3 Months | 4 | 3 | 7 | 14
  Past 4-6 Months | 7 | 3 | 7 | 17
  Past 7-12 Months | 3 | 2 | 2 | 7
  Over 12 Months | 16 | 5 | 17 | 38
Cancer Site [Count of Participants; unit: Participants]
  Lung | 11 | 4 | 11 | 26
  Head and Neck | 20 | 5 | 8 | 33
  Breast | 7 | 0 | 6 | 13
  Gastrointestinal | 5 | 5 | 11 | 21
  Thyroid | 0 | 0 | 2 | 2
  Genitourinary | 3 | 2 | 7 | 12
  Gynecologic | 2 | 2 | 1 | 5
  Bone | 3 | 2 | 4 | 9
  Brain | 1 | 2 | 4 | 7
  Hematologic/Blood | 4 | 4 | 3 | 11
  Other | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Smoking 7-Day Point Prevalence at 12 Weeks
Description: Using intent-to-treat analysis, 3 (7.7%) PhoneQuit, 2 (5.4%) SmartQuit, and 2 (14.3%) GroupQuit patients reported 7-day point prevalence abstinence from smoking. Smart Quit abstinence was verified with CO readings.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline
Number analyzed (Participants) | 37 | 14 | 39
Participants | 2 | 2 | 3

2. Primary Outcome: Reach
Description: Number of smokers visiting the clinics who are enrolled divided by the total number of smokers visiting the clinics.
Time Frame: 12 weeks
Population: Smokers visiting the clinic during the study period
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Smokers visiting the clinic during the study period
Arm/Group | Eligible Patients
Number analyzed (Participants) | 545
Participants | 90

3. Primary Outcome: Treatment Utilization
Description: Percent of enrolled patient who completed any tobacco-use treatment.
Time Frame: 12 weeks
Population: Participants that completed follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline
Number analyzed (Participants) | 12 | 5 | 18
Participants | 7 | 3 | 9

4. Primary Outcome: Mean Treatment Acceptability Score
Description: Treatment Acceptability (TAQ) consisted of 16 items scored on a 0 to 10 scale (0=worst, 10=best). The questions assessed aspects of treatment acceptability, such as helpfulness in reducing smoking and thoughts and feelings related to the treatment. Data represents the mean score across all items (range 0-10).
Time Frame: 12 weeks
Population: Participants who completed tobacco-use treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline
Number analyzed (Participants) | 4 | 2 | 11
score on a scale | 8.1 (1.2) | 5.7 (3.5) | 5.9 (1.8)

5. Secondary Outcome: Change in Cigarettes Smoked Per Day
Description: Change in Mean Cigarettes Smoked Per Day
Time Frame: Baseline to 12 weeks
Population: Participants completing 12 week follow up.
Measure: Mean (Standard Deviation); unit: cigarettes smoked per day
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline
Number analyzed (Participants) | 12 | 5 | 18
cigarettes smoked per day | -4.7 (13.7) | -12.3 (7.5) | -5.0 (6.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Cognitive Behavior Therapy With NRT | Referral to Area Health Education Center | Referral to Qutiline
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/14 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/14 | 0/39
Other Adverse Events (participants affected / at risk) | 0/37 | 0/14 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03482583/Prot_SAP_001.pdf